CLINICAL TRIAL: NCT03168503
Title: Randomised, Double-blind, Placebo Controlled Cross-over Study to Determine the Beneficial Effects of Synbiotics and PromitorTM (Soluble Corn Flour)on Metabolism and Immunity in Healthy 60-80 Years Old Individuals
Brief Title: Synbiotic Approach to Immunity and Metabolism in the Elderly Study
Acronym: SAIMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Health Sciences Research Centre, Life Science Department, University of Roehampton
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC14/06
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Investigator,Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LGG+Promitor™ (Experimental): LGG:10^12 CFU/g Lactobacillus rhamnosus GG (commercialised as LGG) combined with Promitor™:12g fibres/delivered of Soluble Corn Fibre (SCF) as dry powders to be consumed as 250 ml beverages at breakfast.
  Interventions: Dietary Supplement: LGG+Promitor™
- Promitor™ (Experimental): Promitor™:12g fibres/delivered of Soluble Corn Fibre (SCF) as dry powders to be consumed as 250 ml beverages at breakfast.
  Interventions: Dietary Supplement: Promitor™
- LGG-PB12+Promitor™ (Experimental): LGG-PB12:10^12 CFU/g of a pilus-less derivative L. rhamnosus GG combined with Promitor™:12g fibres/delivered of Soluble Corn Fibre (SCF) as dry powders to be consumed as 250 ml beverages at breakfast.
  Interventions: Dietary Supplement: LGG-PB12+Promitor™
- Maltodextrin (Placebo Comparator): Maltodextrin (an oligosaccharide without prebiotic effect) 12g delivered and served as dry powders to be consumed as 250 ml beverages at breakfast.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: LGG+Promitor™ — synbiotic
  Arms: LGG+Promitor™
Dietary Supplement: Promitor™ — Soluble Corn Fiber
  Arms: Promitor™
Dietary Supplement: LGG-PB12+Promitor™ — synbiotic
  Arms: LGG-PB12+Promitor™
Dietary Supplement: Maltodextrin — Control
  Arms: Maltodextrin

SUMMARY:
The aging process leads to a marked decline in immune function (immunosenescence), causing a significant reduction in immune response after vaccination or infections. Dietary intervention is an attractive, safe and non-invasive way to impact on gut bacteria and subsequently the functioning of the immune system. The ability of the dietary supplementation to alter these functions can be of particular importance in those groups that have an underdeveloped, poorly functioning immune system such as infants, immuno-compromised subjects or elderly. Research over the past two decades has provided evidence that administration of probiotics (live microorganisms which, when administered in adequate amounts, confer a health benefit on the host) could enhance immune function. Lactobacilli and bifidobacteria are the most common probiotics used in humans and various strains have been shown to have immunostimulatory properties in vitro and in experimental models, these properties include modulation of cytokine production. evidence exists of the immunostimulating effects of certain probiotics and the potential to use prebiotics to increase the levels of beneficial bacteria (which are known to be reduced in elderly population). Furthermore, by providing a probiotic at the same time as a prebiotic conditions for survival are enhanced. To date, only a small number of studies conducted have been randomised and/or placebo controlled to unequivocally demonstrate efficacies.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of probiotic Lactobacillus rhamnosus GG (commercialised as LGG), a pilus-less derivative L. rhamnosus GG (LGG-PB12)combined with a putative prebiotic PromitorTM (soluble corn fiber) i.e. a synbiotics and PromitorTM (SCF alone) on the faecal microbiota composition, metabolism and immunity in healthy individuals aged 60-80 years.

It consists of a 3 week randomised intervention treatment periods with the synbiotics, prebiotic and placebo control. Any adverse medical events which occur during the trial (e.g. headache, gut symptoms) should be recorded in a diary along with medication taken.

ELIGIBILITY:
Inclusion criteria:

* aged between 60 and 80 years of age.
* in good general health, defined as no comorbidities requiring regular medical follow up
* Ability to communicate well with the investigator and to comply with the requirements of the entire study

Exclusion criteria:

* History or evidence of organic disease of the gastrointestinal tract; such as tumour, irritable bowel syndrome, etc., within the previous 5 years
* Consumed probiotic or prebiotic preparations on a regular basis (at least 3 times per week) in the last 2 weeks and during the trial period
* Former participation in another study involving prebiotic or probiotic preparations or investigational drugs within the previous 6 months, or intention to use such drugs during the course of the study
* Undergone surgical resection of any part of the bowel
* History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma).
* Currently prescribed immunosuppressive drugs
* Intention to use regularly other medication which affects gastrointestinal motility and/or perception
* Current or recent history (within 12 months) of significant drug or alcohol abuse or dependence

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The modulation of the gut microbiota by synbiotics and PromitorTM inflammatory/immune biomarkers | Changes from baseline to 21 days synbiotics and PromitorTM treatment
  Fecal16S rRNA amplicon sequencing to assess changes in fecal bacterial abundance and species diversity

SECONDARY OUTCOMES:
The modulation of immune function by synbiotics and PromitorTM | Changes from baseline to 21 days synbiotics and PromitorTM treatment
  Blood samples analysis to assess changes in cytokines production

OTHER OUTCOMES:
Digestive symptoms | Changes from baseline to 21 days synbiotics and PromitorTM treatment
  Bristol diary form
Microbiota activity (intestinal gas production) | Changes from baseline to 21 days synbiotics and PromitorTM treatment
  Intestinal gas evacuation on standardized diet

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R Gibson, Study Director — The University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No